CLINICAL TRIAL: NCT04996069
Title: Exploratory Study on Effect of Whitening Agent With Emulsion Gel in Xerostomic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Mabi Singh, Associate Professor, Diagnostic Sciences, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001757
Record Dates: First submitted 2021-07-29; First posted 2021-08-09 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: * Primary aim: To see a reduction in the self-reported subjective perception of dryness in the oral cavity.
  * Secondary aims: To measure self-reported sensitivity of the teeth, self-reported perception of teeth whiteness, and objective measurement of improvement of saliva production.
Masking Description: This will be an open label study; thus no randomization plan is necessary.There will be no blinding for this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): This is a single arm study. All subjects enrolled will be apart of the experimental group. Subjects in this group will use Crest Whitening Emulsions on their teeth up to 4 times a day for 7 days in order for the study team to evaluate if the study intervention product increases saliva production in this Xerostomic population.
  Interventions: Device: Crest Whitening Emulsions

INTERVENTIONS:
Device: Crest Whitening Emulsions — Subjects with Xerostomia will be asked to apply the study intervention product to their teeth up to 4 times per day for 1 week to investigate if the study intervention product increases saliva production in this dry mouth populaiton.

SUMMARY:
Xerostomia, is a subjective sensation of dryness of the mouth. There are more than 700 medications that can lead to the salivary hypofunction that results in dry mouth. This study will investigate a semi solid cohesive gel (referred to as Whitening Gel) that has the primary marketed purpose of teeth whitening. We theorize that the whitening gel's retention in the oral cavity is longer than rinse forms and this is likely to promote the flow of saliva by stimulating taste buds which could alleviate the sensation of dryness in the oral cavity. This will be a single center, two visit study investigating the effectiveness of dryness in the oral cavity, whiteness of teeth, and teeth sensitivity after one week's use of whitening agent.

DETAILED DESCRIPTION:
Aims:

* Primary aim: To see a reduction in the self-reported subjective perception of dryness in the oral cavity.
* Secondary aims: To measure self-reported sensitivity of the teeth,. self-reported perception of teeth whiteness, and objective measurement of improvement of saliva production.

Background and Rationale:

Xerostomia, is a subjective sensation of dryness of the mouth, which may have a significant effect in a persons quality of life. The sensation of dryness of the mouth may be caused by autoimmune diseases which attack the saliva producing glands irreversibly e.g., salivary glands, or the sensation of dryness could be caused by therapeutic radiation, which can destroy the salivary glands at the genetic level and impede their functions. Additionally, there are more than 700 medications including antihypertensives, anti-anxiety agents, psychiatric remedies, and antihistamines that can effect neural transmission. Neural transmission is when the neuro transmission is hindered reversibly leading to the salivary hypofunction that results in dry mouth. It is estimated that 12-47% of the elderly and 10-19.3% in their early 30's suffer from dry mouth (Thomson et al 2005)(Guggenheimer et al 2003). In a study, it was found that the prevalence of xerostomia was 10.0% (with no apparent gender difference) among 32-year-olds and was significantly higher among those taking antidepressants (odds ratio =4.7) (Murray et al 2006). At risk groups may present much higher (60+%) rates of xerostomia. A systemic literature review suggests a prevalence of 27 -32% of the medicated population suffer from xerostomia as a side effect (Guggenheimer et al 2003).

Saliva, the bulk fluid of the oral cavity is very important in maintaining the functions and balance in the oral cavity including candidiasis and enamel erosion prevention. In past studies, residual mucosal fluid levels were seen to vary in different oral cavity sites from an average of 70-100 μm (Collins et al 1987)(Pramanik et al 2010). In addition, the vault of the hard palate has much less mucosal fluid thickness than the floor of the mouth. Over the moisture layer is the lipid layer and reduction or loss of this moisture layer can contribute to the subjective perception of the dryness in the mouth. An addition of the lipid layer will also increase lubrication in the oral cavity.

Unstimulated salivary flow in dry mouth patients has shown an increased clinical oral dryness score and mucosal wetness is at a significantly reduced rate (p<0.05) when compared with healthy subjects (Osailan et al 2010).

Historically, various products containing methylcellulose, water, oily emulsions etc., have been used to alleviate the subjective sensation of dryness in the oral cavity in the forms of rinse, gel, ointment and paste. However, the alleviation of the dry mouth symptoms has been varied.

The study product contains an inert hydrophobic phase in an amount from 30% to 98%, preferably from 40% to 90% by weight of the composition. It also contains an emulsifying system in an amount from 1% to 10%, preferably from 3% to 7% by weight of the composition.

P&G's whitening gel emulsifying system is comprised of at least one surfactant having an hydrophilic-lipophilic balance (HLB) <10, preferably comprised between 3 and 7, and at least one surfactant with HLB>10, preferably comprised between 12 and 16.

The optimal duration and frequency of application for whitening is up to 4 times a day. For the purpose of this study, the whitening gel will set on the subject's teeth for 5 minutes during each use.

The product being used is a commercially available product, known as "Crest Whitening Emulsions", will be used as the investigative product. There will be no active control group. This is not the first time the P&G whitening gel will be used in humans. We do believe this is the first study investigating dry mouth sensation from using a whitening gel.

The amount of each dose should be enough to cover the entire tip of the whitening wand, approximately ½ a tsp. The use of the study product in this study will be for what they are approved for. Per the manufacturer's instructions, study subjects will be asked to apply the study product up to 4 times a day.

Study Procedures

Visit 1 (1-1.5 hours) Screening/ Baseline (Day 0)

1. Subject will be called 1-2 days before their appointment to confirm that in order to participate, they must:

   1. Not consume alcohol for 24 hours prior to their visit.
   2. Not brush their teeth for 1.5 hours prior to their visit.
   3. Not have had anything to eat or drink (including chewing gum or eating candy) for 1.5 hours prior to their visit). Water is acceptable to drink up to 1 hour prior to the study visit.
   4. Not smoke 1.5 hours prior to their visit.
2. The subjects will be asked to read the informed consent form (ICF). Subjects will be given ample time to have any questions answered. If a subject decides to participate, he or she will be asked to sign the ICF. A copy of the ICF will be given to the subject.
3. Subject will be asked to complete demographic information and a medical history.
4. An oral exam, including evaluation of oral cavity, soft and hard tissues, will be completed following standard of care procedures in US dentistry using a mouth mirror and dental explorer.
5. Subject medications with potential side effects being dry mouth will be verified using the Physician's Reference Desk.
6. Saliva Collection 1 (pre-product application): Saliva will be collected by asking subjects to do nothing but drool into a pre-weighed vial for 5 minutes (referred to as the Drooling Method). The post collection weight will be subtracted from the pre-weight to determine the flow rate. The saliva samples will be discarded after they are weighed.
7. A paper questionnaire will be given to subject to complete before application of study product and after application of study product. Questionnaire includes Visual Analogue Scale (VAS) questionnaire on dry mouth, quantity of saliva, and perceived sensitivity of teeth.
8. Inclusion/exclusion criteria will be evaluated and eligibility for the study will be determined.
9. Demonstration and application of study product:

   a. A visual and oral demonstration of application of the whitening gel will be performed by a study team member. The script for the demonstration will be the one provided in the information packet in each study product box so the subject can bring the instructions home. The study team member will mimic the necessary steps to properly apply the gel, without using the product. The study team member will then have the subject complete the steps while applying the gel to their own teeth. Subjects will then be asked to sit for 5 minutes to let the gel set on their teeth. During that time, the subject can fill out the post-application questionnaire.
10. Saliva Collection 2 (post-product application): Saliva will be collected using the same Drooling Method as Saliva Collection 1. The saliva samples will be discarded after they are weighed.
11. Photographs of subject teeth will be taken by a standard dental camera. The photos will only contain subject teeth and oral cavity with no subject identifiers visible. In addition to the ICF, the subjects will be asked to sign a photo release form. If the subject does not wish to sign this form, their photographs will not be taken. Those who do not consent to having their photos taken will be tracked in the enrollment log
12. Distribution of study product and diary: One box of study whitening gel product, (0.88Oz) toothpaste, and a toothbrush will be dispensed by study team members. This is to ensure all participants are using the exact same dental products during the trial period. The subjects will be asked to not use any other oral tools or products during the trial period aside from the ones distributed by the study team at Visit 1. A diary will also be dispensed for the record keeping of the application of the products. A study team member will again verbally tell the participant the instructions that are provided with the study product and that per the instructions, they can apply the product up to 4 times per day until their next study visit. The same script from step 9.a. will be used.
13. Gift card will be distributed upon successful completion of visit.

Visit 2 (1-1.5 hours) Final Visit - 7 ∓ 2 days after visit 1

1. Subject will be called 1-2 days before their appointment to confirm that in order to participate, they must:

   1. Not consume alcohol for 24 hours prior to their visit.
   2. Not brush their teeth for 1.5 hours prior to their visit.
   3. Not have had anything to eat or drink (including chewing gum or eating candy) for 1.5 hours prior to their visit). Water is acceptable to drink up to 1 hour prior to the study visit.
   4. Not smoke 1.5 hours prior to their visit.
2. Medical history will be reviewed, and any changes will be noted. Any changes to medications will also be reviewed and noted.
3. Eligibility and subject withdrawal criteria will be reviewed to ensure the subject still qualifies for the study.
4. Subject medications with potential side effects being dry mouth will be verified using the Physician's Reference Desk. Subjects will be asked to confirm that they have taken their medications as prescribed since Visit 1.
5. An oral exam, including evaluation of oral cavity, soft and hard tissues, will be completed following standard of care procedures in US dentistry using a mouth mirror and dental explorer.
6. Saliva Collection 1 (pre-product application): Saliva will be collected using the drooling method for 5 minutes into a pre-weighed vial. The post collection weight will be subtracted from the pre-weight to determine the flow rate. The saliva samples will be discarded after they are weighed.
7. The paper questionnaire will be given to subject to complete before application of study product and after application of study product. The questionnaire includes the Visual Analogue Scale (VAS) questionnaire on dry mouth, quantity of saliva, and perceived sensitivity of teeth.
8. Application of study product: A study team member will ask the subjects to apply the gel to their teeth. Subjects will then be asked to sit for 5 minutes to allow the gel to set on their teeth. During that time, subjects will fill out the post- application questionnaire.
9. Saliva Collection 2 (post-product application): Saliva will be collected using the same drooling method as Saliva Collection 1. The saliva samples will be discarded after they are weighed.
10. Photographs of subject teeth will be taken by a standard dental camera. The photos will only contain subject teeth and oral cavity with no subject identifiers visible.
11. The study diary and any leftover product will be collected.
12. Gift card will be distributed upon successful completion of visit.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* The inability to produce more than 0.18mL/min of unstimulated saliva.
* Score of 5 or more in the VAS dry mouth scale, evaluated in the mouth feel questionnaire.
* Evidence of currently taking Xerostomia-inducing medication such as, antihypertensives, anti-anxiety agents, psychiatric remedies, antihistamines.
* Subject not currently using any teeth whitening or desensitizing products that contain potassium nitrate such as Sensodyne or Pronamel.
* Subject willing to comply with the study regimen and products.

Exclusion Criteria

* Subjects who are currently pregnant (self-reported).
* Subjects able to produce more than 0.18mL/min of unstimulated saliva
* Subjects that have ever received therapeutic radiation in the head and neck area.
* Subjects with a diagnosis of conditions that would affect salivary flow such as Sjogren's Syndrome.
* Subjects with a condition the investigator believes not suitable for the study such as autoimmune diseases that impact salivary flow.
* Subjects that currently use whitening toothpaste, desensitizing toothpaste, or any other products causing similar results.
* Subjects currently participating in any other research studies.
* Subject unable to provide consent (ex. Cognitively impaired adults).
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mabi Singh, DMD, MS, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Apperley O, Medlicott N, Rich A, Hanning S, Huckabee ML. A clinical trial of a novel emulsion for potential use as a saliva substitute in patients with radiation-induced xerostomia. J Oral Rehabil. 2017 Nov;44(11):889-895. doi: 10.1111/joor.12545. Epub 2017 Aug 20. PMID 28741683
- [Background] Collins LM, Dawes C. The surface area of the adult human mouth and thickness of the salivary film covering the teeth and oral mucosa. J Dent Res. 1987 Aug;66(8):1300-2. doi: 10.1177/00220345870660080201. PMID 3476596
- [Background] Pramanik R, Osailan SM, Challacombe SJ, Urquhart D, Proctor GB. Protein and mucin retention on oral mucosal surfaces in dry mouth patients. Eur J Oral Sci. 2010 Jun;118(3):245-53. doi: 10.1111/j.1600-0722.2010.00728.x. PMID 20572857
- [Background] Osailan S, Pramanik R, Shirodaria S, Challacombe SJ, Proctor GB. Investigating the relationship between hyposalivation and mucosal wetness. Oral Dis. 2011 Jan;17(1):109-14. doi: 10.1111/j.1601-0825.2010.01715.x. Epub 2010 Oct 28. PMID 21029258
- [Background] Murray Thomson W, Poulton R, Mark Broadbent J, Al-Kubaisy S. Xerostomia and medications among 32-year-olds. Acta Odontol Scand. 2006 Aug;64(4):249-54. doi: 10.1080/00016350600633243. PMID 16829502
- [Background] Thomson WM. Issues in the epidemiological investigation of dry mouth. Gerodontology. 2005 Jun;22(2):65-76. doi: 10.1111/j.1741-2358.2005.00058.x. PMID 15934347
- [Background] Guggenheimer J, Moore PA. Xerostomia: etiology, recognition and treatment. J Am Dent Assoc. 2003 Jan;134(1):61-9; quiz 118-9. doi: 10.14219/jada.archive.2003.0018. PMID 12555958

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 25
Completion of the Study | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] — Population: One subject had more unstimulated saliva than .18 ml/min at baseline and was not included in the analysis.
  years | 58 [23 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25
Salivary flow [Mean (Standard Deviation); unit: ml/min] | .067 (.063)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Perception of Mouth Dryness
Description: At both study visits, subjects will be asked to complete a visual analog scale (VAS) before and after the application of the study product to establish a self-reported subjective perception of the oral cavity. The scale ranges from 0 to 10 and the higher the score indicates the more Xerostomic the subject.
Time Frame: visit 1 and visit 2 pre and post product application on Day 1 and day 7
Population: unstimulated salivary flow below 0.18 ml/min at the baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Exploratory Study on Effect of Whitening (Agent) With Emulsion on Xerostomic Population.: medication induced xerostomic population with unstimulated salivary flow below 0.18ml/min
- Second/Final Visit +/- 7 Days: The same as visit one and pre questions
Arm/Group | Exploratory Study on Effect of Whitening (Agent) With Emulsion on Xerostomic Population. | Second/Final Visit +/- 7 Days
Number analyzed (Participants) | 24 | 24
units on a scale
  Subjective perception prior to product application | 6.92 (1.53) | 6.46 (2.62)
  Subjective perception after the product application | 4.21 (2.50) | 3.46 (2.54)
Statistical Analysis 1: Comparison: Exploratory Study on Effect of Whitening (Agent) With Emulsion on Xerostomic Population. vs Second/Final Visit +/- 7 Days; Test type: Superiority — No power calculation performed; p = .45, t-test, 2 sided — p value threshold is .05

2. Secondary Outcome: Change in Saliva Production Measured in ml/Min
Description: For the objective measurement of the improvement of the saliva production; subjects will be asked to drool into a pre-weighed vial for 5 minutes before application of the study product and again after application at both visits. The difference in weight will be calculated to evaluate what effectiveness the study product may have in saliva production
Time Frame: visit 1 and visit 2 pre and post saliva production in day 1 and day 7
Measure: Median (Standard Deviation); unit: mL/Min
Arm/Group | All Participants
Number analyzed (Participants) | 24
mL/Min
  Pre product application salivary flow (Day 1) ml/min | 0.06 (0.08)
  Post product application salivary flow (Day 1) ml/min | 0.19 (0.08)
  Pre product application salivary flow (Day 7) ml/min | 0.14 (0.21)
  Post product application salivary flow (Day 7) ml/min | 0.21 (0.33)

3. Secondary Outcome: Perceived Sensitivity of Teeth Between Visit 1 and 2
Description: At both study visits, subjects will be asked to complete a visual analog scale to establish if there is a difference between self-reported sensitivity. The scale ranges from 0 to 10 and the higher the score indicates the more sensitive the subject's teeth.
Time Frame: 7 days between visit 1 and visit 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exploratory Study on Effect of Whitening (Agent) With Emulsion on Xerostomic Population. | Second/Final Visit +/- 7 Days
Number analyzed (Participants) | 24 | 24
units on a scale
  Pre product application (sensitivity of teeth) | 3.61 (3.46) | 3.72 (3.33)
  Post Product application (sensitivity of teeth) | 2.30 (3.14) | 1.56 (2.7)

ADVERSE EVENTS:
Time Frame: The duration of the study - about 6 months.
Description: The definition of adverse event and serious adverse event, used to collect adverse event information, does not differ from the clinicaltrials.gov Definitions
Groups:
- All Participants: No adverse reaction were noted.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT04996069/Prot_SAP_000.pdf